CLINICAL TRIAL: NCT02773277
Title: Prospective Assessment of Peripheral-vestibular Function After Skull Base Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: vHIT_surgery
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Vestibular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single intervention arm (Experimental): All patients will be assigned the intervention arm and will receive head-impulse testing before and in the days after skull base surgery.
  Interventions: Other: head-impulse testing

INTERVENTIONS:
Other: head-impulse testing — all patients will receive quantitative head impulse testing using video goggles for all six semicircular canals.

SUMMARY:
Due to its localization in the cerebello-pontine angle, the vestibulo-cochlear nerve is at risk to damage during surgery performed nearby. In most cases, peripheral-cochleovestibular hypofunction recovers over the following weeks as the mechanism of damage is rather demyelination than axonal damage. The rate, intensity and extent of recovery of such perioperative peripheral-vestibular damage is not known.

DETAILED DESCRIPTION:
Due to its localization in the cerebello-pontine angle, the vestibulo-cochlear nerve is at risk to damage during surgery performed nearby, e.g. when removing an epidermoid cyst, treating a neuro-vascular conflict of the trigeminal nerve or resecting a petroclival meningeoma. Intense vertigo and dizziness accompanied by spontaneous nystagmus following Alexander's law, nausea and gait imbalance may be noted in these patients along with cochlear hypofunction (hearing loss). In most cases, peripheral-cochleovestibular hypofunction recovers over the following weeks as the mechanism of damage is rather demyelination than axonal damage. The rate, intensity and extent of recovery of such perioperative peripheral-vestibular damage is not known. Besides peripheral-vestibular hypofunction, transient cerebellar hypofunction may arise, presenting with similar complaints (vertigo, nausea, gait imbalance), however, distinct subtle ocular motor findings.

The aim of this study is to characterize the frequency and pattern of iatrogenic peripheral-vestibular and cochlear hypofunction and to follow-up on the speed and extent of recovery. The investigators hypothesize that peripheral-vestibular and cochlear damage may be observed in a significant fraction of neurosurgical treatments in the posterior fossa including the cerebello-pontine angle. While initially deficits may be major, recovery is expected to be substantial or even complete due to peripheral restoration. As an important differential diagnosis, the investigators will evaluate also for potential (transient) cerebellar loss of function.

In order to quantify peripheral-vestibular function the investigators will use a CE-certified videooculography device to record responses to the head-impulse test before and in the days following elective skull base surgery. the video-head impulse test (vHIT) allows a quantitative video-based assessment of the functional integrity of all semicircular canals (MacDougall et al. 2013). By use of a high-speed video-camera mounted on goggles this test quantifies the vestibulo-ocular reflex (VOR), which is the fastest human reflex and allows the recognition and visual fixation of objects while head turns or ambulation. This test is used on a routine basis in our clinic and includes brief and fast, but small amplitude head turns (10-15° excursion) in the planes of the different semi-circular canals (SCCs). The SCCs are tested in three pairs in the horizontal, RALP (right anterior, left posterior) and LARP (left anterior, right posterior) plane (Weber et al. 2008). During testing the participant is asked to fixate a visual target straight ahead. Duration of this test: about 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older
2. informed consent
3. absence of exclusion criteria

Exclusion Criteria:

1. peripheral-vestibular deficit before surgery
2. disturbed consciousness
3. diagnosis of vestibular schwannoma
4. other neurological or systemic disorder which can cause dementia or cognitive dysfunction
5. known neck pain or status post neck trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
gain of the angular vestibulo-ocular reflex | comparison before surgery and up to 30 days post surgery
  in all patients the mean gain for each semicircular canal will be determined
Cumulative saccade amplitudes per trial [°/trial] of the angular vestibulo-ocular reflex | comparison before surgery and up to 30 days post surgery
  in all patients the cumulative saccade amplitudes per trial for each semicircular canal will be determined

SECONDARY OUTCOMES:
clinical testing of the horizontal head-impulse test | comparison before surgery and up to 30 days post surgery
  besides the vHIT, patients will be examined clinically, including testing for central-type acute vestibular syndrome.
clinical testing for gaze-evoked nystagmus | comparison before surgery and up to 30 days post surgery
  besides the vHIT, patients will be examined clinically, including testing for central-type acute vestibular syndrome.
clinical testing for skew deviation by use of the alternating cover test | comparison before surgery and up to 30 days post surgery
  besides the vHIT, patients will be examined clinically, including testing for central-type acute vestibular syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Krayenbühl, MD, Principal Investigator — University Hospital Zurich, Neurology

IPD SHARING:
Plan to Share IPD: No